CLINICAL TRIAL: NCT03820297
Title: Effects Of Anti-Stigma Intervention For Chinese American Older Adults With Mood And Anxiety Disorders
Brief Title: Anti-stigma Intervention for Chinese American Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Substance Abuse and Mental Health Services Administration (SAMHSA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-01236
Record Dates: First submitted 2019-01-25; First posted 2019-01-29 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Mood Disorders; Anxiety Disorders
MeSH Terms: conditions — Mood Disorders; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anti-Stigma Group (Other): Complete a 10 weekly anti-stigma group intervention (ASGI) in addition to several self-report internalized stigma and psychiatric measures.
  Interventions: Behavioral: 10 sessions of ASGI

INTERVENTIONS:
Behavioral: 10 sessions of ASGI — 10-session intervention will occur weekly for 45 minutes per session: psychoeducation about mood and anxiety disorders, focusing on identification of risk factors and biological theory to counter stigma; psychoeducation regarding 'therapeutic modules' (psychotropics and psychotherapy) to treat depression, with an emphasis on the importance of psychiatric treatment adherence, providing behavioral strategies for anticipated and experienced forms of mental illness related work, social, or family discrimination

SUMMARY:
Approximately 50 participants will be enrolled and screened to achieve 45 eligible patients with mood/anxiety disorders to complete a 10 weekly anti-stigma group intervention (ASGI) in addition to several self-report internalized stigma and psychiatric measures.This study will examine changes in internalized stigma and psychiatric symptoms pre- and post-ASGI with 3 months post-intervention follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported Chinese heritage;
* 55 years or older
* Mandarin and/or Cantonese speaking and ability to read and/or comprehend spoken Chinese language.
* Currently receiving treatment from a mental health provider at Gouverneur Medical Center Asian Bicultural Clinic (GMC ABC) and willing to continue mental health care through the study.
* Willing to provide release for communication between primary mental health care provider and study staff throughout the study.
* Documented by mental health provider after consent for release of information as having mood and anxiety disorder diagnosis in the past year;
* A willingness to participate in the ASGI with stated availability;
* Able and willing to provide informed consent.

Exclusion Criteria:

* Lifetime psychosis, neurocognitive, or significant neurological disorders;
* Current manic episode;
* Past 6 months of alcohol/substance use disorder;
* Serious safety concerns of suicide or homicide.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-08-19 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
Self stigma of mental illness scale | 23 weeks
  This 40-item self-report scale assesses the extent of patient self-stigma. Items are rated on a 9-point Likert-type scale (1= Strongly Disagree; 9= Strongly Agree).
  Total score from 1 to 9 (average score) Higher score means worse outcome
Recovery assessment scale | 23 weeks
  Empowerment will be assessed using the 15-item scale from the Recovery Assessment Scale. This scale measures domains of recovery including 1) personal confidence and hope 2) willingness to ask for help 3) goal and success orientation 4) reliance on others 5) symptom coping. Patients are asked to describe themselves using a 5-point agreement scale (1= strongly disagree, 5= strongly agree) regarding their recovery.
  Total score from15 to 75 (summed score) Higher score means better outcome
Self-protective Withdrawal and Secrecy scale | 23 weeks
  Changes in use of self-protective withdrawal and secrecy as a strategy for coping with public stigma will be evaluated using two scales to assess patients' responses to their stigmatized status.
  1. Secrecy subscale: a 5-item Likert-type scale (1=strongly agree, 6=strongly disagree) assessing use of concealment of mental illness.
     Total score: 5 to 30 (summed score)
  2. Withdrawal subscale consists of 7 items (1=strongly agree, 6=strongly disagree) assessing "limiting social interaction to those who know about and tend to accept one's stigmatized condition".
  Total score: 6 to 42 (average score).
  For the overall scale, summed score will be used. Higher score means better outcome

SECONDARY OUTCOMES:
Changes in social support | 23 weeks
  The subjective support and social interaction subscales from the Abbreviated Duke Social Support Scale (ADSSS) will be used to measure changes in social support. It is an 11-item Likert-type scalewhich has been shown to correlate well with mental and physical health outcomes.
  1. Social interaction sub-scale: patients are asked 4 items to describe their telephone and face-to-face interaction patterns during the past week (1=none, 2=1-2 people, 3=more than 2 people).
     Total score: 4 to 12 (summed score ).
  2. Satisfaction with social support sub-scale: they are asked to respond to 7 questions such as "Does it seem that your family and friends understand you most of the time, some of the time, or hardly ever?" (1=hardly ever, 2=some of the time, 3=most of the time).
  Total score: 7 to 21 (summed score)
  For the overall scale, total score from 11 to 33 (summed score of two subscales). A higher score means better outcome
Changes in patient depressive symptoms measured by Patient Health Questionnaire-9 (PHQ-9) | 23 weeks
  The Patient Health Questionnaire-9 (PHQ-9) is a 9-item interview assessing depressive symptoms which is a reliable and valid measure of depression severity (0=not at all, 1=several days, 2=more than half the days, 3=nearly everyday).
  Total score: 27 (summed score). A higher score means worse outcome
Changes in patient anxiety symptoms associated with stigma reduction | 23 weeks
  The Generalized Anxiety Disorder 7-item Scale (GAD-7) is a 7-item interview assessing anxiety symptoms (0=not at all, 1=several days, 2=more than half the days, 3=nearly everyday).
  Total score: 21 (summed score will be used). A higher score means worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Simon, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States